CLINICAL TRIAL: NCT06256744
Title: Resistance Exercise-induced Anabolism in Youths and Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Bareket Falk, Professor, Brock University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BFalk
Record Dates: First submitted 2023-12-28; First posted 2024-02-13 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Dietary Supplementation; Exercise
Keywords: Children; Muscle; Protein; Resistance training
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: children, adolescents and adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein supplementation (Experimental): Protein supplementation
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Resistance exercise

SUMMARY:
Resistance exercise training (RET) in children and adolescents has become a popular area of research, with a growing body of evidence supporting its use. Position and consensus statements about RET for children indicate that it is safe and effective at increasing muscular strength, improving sport performance, and mitigating injury risk. Neural and muscular mechanisms can improve muscle strength following RET. Neural factors include improved recruitment and firing of an individual's motor units, and muscular factors primarily include an increase in the size of the muscle (hypertrophy).

In children, little is known about how these mechanisms relate to muscle strength. There is very little evidence of morphological changes following RET in children. Therefore, conventional wisdom is that children rely only on neural factors to improve strength following RET. Nevertheless, some studies have suggested RET-induced muscle hypertrophy in children and adolescents, indicating that with certain training protocols, children may achieve muscle growth.

Hypertrophy of muscle fibres occurs when the rate of muscle protein synthesis (MPS) is greater than the rate of protein breakdown, and is enhanced with the ingestion of dietary amino acids. Due to ethical concerns with obtaining muscle samples (i.e., from muscle biopsies) in pediatric populations, MPS rates have not been previously assessed following RET in children. Recent advancements in stable-isotope methodology (specifically, leucine) allow for the estimation of MPS in a non-invasive breath test.

The objective of the proposed research is to examine the effects of an acute bout of RET on leucine retention (a proxy for MPS) in children, adolescents, and adults using a non-invasive breath test.

DETAILED DESCRIPTION:
Resistance exercise training (RET) in children and adolescents has become a popular area of research, with a growing body of evidence supporting its use. Position and consensus statements about RET for children indicate that it is safe and effective at increasing muscular strength, improving sport performance, and mitigating injury risk. Neural and muscular mechanisms can improve muscle strength following RET. Neural factors include improved recruitment and firing of an individual's motor units, and muscular factors primarily include an increase in the size of the muscle (hypertrophy).

In children, little is known about how these mechanisms relate to muscle strength. There is very little evidence of morphological changes following RET in children. Therefore, conventional wisdom is that children rely only on neural factors to improve strength following RET, possibly due to their lower levels of circulating androgens. Nevertheless, some studies have suggested RET-induced muscle hypertrophy in children and adolescents, indicating that with certain training protocols, children may achieve muscle growth.

Hypertrophy of muscle fibres occurs when the rate of muscle protein synthesis (MPS) is greater than the rate of protein breakdown, and is enhanced with the ingestion of dietary amino acids. Due to ethical concerns with obtaining muscle samples (i.e., from muscle biopsies) in pediatric populations, MPS rates have not been previously assessed following RET in children. Recent advancements in stable-isotope methodology allow for the estimation of MPS in a non-invasive breath test, which is based on the retention of an essential amino acid (i.e., leucine) that is preferentially metabolized within skeletal muscle. Given that amino acids can only be 'stored' in functional body proteins with any excess being converted to energy (i.e., oxidized), this non-invasive technique is ideal to safely estimate the anabolic (i.e., growth) potential of RET in children. Indeed, similar techniques using ingested stable isotopes have been safely and successfully used in children and adolescents.

The objective of the proposed research is to examine the effects of an acute bout of RET on leucine retention (a proxy for MPS) in children, adolescents, and adults using a non-invasive breath test. It is hypothesized that following a bout of RET, protein retention will be augmented in all groups compared to a non-exercised condition. However, due to a greater basal rate of leucine retention (i.e., for growth processes), the RET-induced increase will be relatively lower in the children and adolescents.

Design: The proposed study will use a cross-sectional design that will compare leucine retention at rest, as well as following a bout of resistance exercise in children, adolescents, and adults.

Procedures: Participants will be required to make three visits to the Applied Physiology Laboratory at Brock University for the completion of all procedures.

During visit 1, the participants and their guardian(s) (if under the age of 18) will be informed of all tests and procedures that will take place over the duration of the study. Written and verbal consent will be obtained from the participants and their guardians (in the case of children and adolescents) before proceeding with further questionnaires. Questionnaires screening for medical concerns, pubertal stage, athletic training practices, menarche and oral contraceptive use (for adolescent and adult females), habitual eating habits, and habitual physical activity will then be completed. Anthropometric measurements will also be performed (i.e., height, seated height, body fat composition, skinfold thickness, limb lengths, limb circumferences, muscle cross sectional area). Following questionnaires and anthropometric measurements, participants will be familiarized with the exercises to be performed in their RET session. Each participant's strength will also be tested for these exercises.

Visits 2 and 3 will serve as the experimental sessions and will consist of a RET and a rest session, done in a counterbalanced order. For these sessions, participants will arrive fasted in the morning, and will be provided with a standardized breakfast and beverage. At the beginning of the experimental sessions, participants will have their breath collected. This will be followed by RET in one of the sessions, or continued rest. A dose of L-[1-13C]leucine isotope will then be consumed based on each participant's body mass (within a protein and carbohydrate beverage) and the breath of each participant will continue to be collected for the next 5 hours (total of 11 breath samples). A small snack will be given to each participant during this breath collection period.

Resistance Exercise: Strength testing and the training protocol will involve the following exercises which will all be performed using strength training machines. The use of such equipment is considered safer than the use of free weights as there are less degrees of freedom during limb movements, preventing technical failure prior to muscular fatigue. The following exercises will be performed: seated leg press, seated overhead press, seated chest press, seated horizontal row. Exercises will be performed with techniques described by the Canadian Society for Exercise Physiology (CSEP - PATH, 2021).

The RET protocol will comprise of 3-5 sets of each exercise at 70-80% of 1RM. Each exercise will be performed until failure (i.e., until the participant can no longer complete the movement with safe technique), as this has been shown to be optimal for stimulating MPS and eliciting muscle hypertrophy. Approximately 8-15 repetitions are expected to be completed per set and ~90s of rest will be given between sets. A similar acute RET protocol has previously been shown to be a sufficient stimulus to elicit differences in leucine retention compared to rest (tested using the non-invasive breath test that will be used in the proposed study) in adults.

The participants in the proposed study will be male and female prepubertal children (~7-12 years), adolescents (~13-16 years), and adults (18-35 years).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* free of injury that would prevent resistance exercise

Exclusion Criteria:

* consumed any medications in the past year which may affect muscle function
* had an injury in the past 6 months that would limit the movements required for the protocols
* been told that has diabetes
* been told that had a heart problem
* been told that have a breathing problem (e.g., asthma)
* been told that sometimes experience seizures
* had joint instability or ongoing join chronic pain
* been told that had kidney problems
* had stomach problems such as ulcers
* experience prolonged bleeding after a cut

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Leucine retention | During the experimental session, expired air is collected pre-ingestion and every 30minutes. i.e., at -60, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes.
  retention is calculated as intake minus leucine in expired air (mg). This test involves blowing into a breath collection bag before, and every ~30 minutes after (for ~300 minutes) ingesting a powdered-amino acid supplement (modeled after egg protein - the WHO/FAO gold standard protein source) mixed with water. The supplement will contain 0.25 g/kg body mass of protein as crystalline amino acids, 0.75 g/kg body mass of carbohydrate (~4kcal/kg of body mass), and will be enriched with 1 mg/kg of L-[1-13C]leucine (Cambridge Isotope Laboratories Inc., Tewksbury, MA, USA), which is a stable isotope that can be detected in the breath of the participants when not used for protein synthesis. The amount of the isotope that is expelled (oxidized) in the breath of the participant can be detected using continuous-flow isotope ratio mass spectrometry (ID-Microbreath; Compact Science Systems, Newcastle, UK), which allows for the estimation of leucine retention (intake - oxidation)

SECONDARY OUTCOMES:
body mass | baseline in each experimental session
  mass in kg
body height | baseline, pre-intervention
  height in cm
arm circumference | baseline in each experimental session
  arm circumference in cm
thigh circumference | baseline in each experimental session
  circumference in cm
Skinfold thickness - triceps | baseline, pre-intervention
  skinfold thickness in mm (using Harpenden calipers)
skinfold thickness - subscapula | baseline, pre-intervention
  skinfold thickness in mm (using Harpenden calipers)
Body composition (BIA) | baseline, pre-intervention
  Bioelectrical impedance analysis (BIA) - percentage of body fat
Muscle thickness - thigh, upper arm | baseline, pre-intervention
  muscle thickness in mm - using ultrasound system
[13C]leucine in urine | baseline and post-each experimental session. i.e., at -60 and 300 minutes
  concentration in microgram, using mass spectrometry
maximal strength (1RM) | baseline, pre-intervention
  maximal weight lifted/pushed in kg - seated leg press, seated overhead press, seated chest press, seated horizontal row
oxygen consumption | During the experimental session, every 30 minutes: i.e., at -60, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes.
  Oxygen consumption (l/min) - using open circuit metabolic system
carbon dioxide production | During the experimental session, every 30 minutes: i.e., at -60, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes. (every 30min)
  carbon dioxide production (l/min) - using open circuit metabolic system
nutritional intake | baseline, pre-intervention
  Nutritional intake (carbohydrates, fats, proteins) - in g/day and as % or daily recommendation. Using Food Frequency questionnaire and 24-h recall.
leisure time physical activity level | baseline, pre-intervention
  physical activity level, using the Godin-Shephard leisure time questionnaire. Minimum score is 0, with no maximum limit. Higher score reflects more physical activity
Pubertal stage (children and adolescents only) | baseline, pre-intervention
  Based on secondary sex characteristics of pubertal hair (Tanner scale). Stages are 1-5, where 1 is pre-pubertal and 5 is post-pubertal

CONTACTS AND LOCATIONS:
Overall Officials: Bareket Falk, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will only be available to researchers directed involved in the study

REFERENCES:
- [Background] Behm DG, Faigenbaum AD, Falk B, Klentrou P. Canadian Society for Exercise Physiology position paper: resistance training in children and adolescents. Appl Physiol Nutr Metab. 2008 Jun;33(3):547-61. doi: 10.1139/H08-020. PMID 18461111
- [Background] Enoka RM. Muscle strength and its development. New perspectives. Sports Med. 1988 Sep;6(3):146-68. doi: 10.2165/00007256-198806030-00003. PMID 3055145
- [Background] Faigenbaum AD, Kraemer WJ, Blimkie CJ, Jeffreys I, Micheli LJ, Nitka M, Rowland TW. Youth resistance training: updated position statement paper from the national strength and conditioning association. J Strength Cond Res. 2009 Aug;23(5 Suppl):S60-79. doi: 10.1519/JSC.0b013e31819df407. PMID 19620931
- [Background] Fukunaga T, Funato K, Ikegawa S. The effects of resistance training on muscle area and strength in prepubescent age. Ann Physiol Anthropol. 1992 May;11(3):357-64. doi: 10.2114/ahs1983.11.357. PMID 1642736
- [Background] Granacher U, Goesele A, Roggo K, Wischer T, Fischer S, Zuerny C, Gollhofer A, Kriemler S. Effects and mechanisms of strength training in children. Int J Sports Med. 2011 May;32(5):357-64. doi: 10.1055/s-0031-1271677. Epub 2011 Mar 4. PMID 21380967
- [Background] Lim C, Nunes EA, Currier BS, McLeod JC, Thomas ACQ, Phillips SM. An Evidence-Based Narrative Review of Mechanisms of Resistance Exercise-Induced Human Skeletal Muscle Hypertrophy. Med Sci Sports Exerc. 2022 Sep 1;54(9):1546-1559. doi: 10.1249/MSS.0000000000002929. Epub 2022 Apr 6. PMID 35389932
- [Background] Lloyd RS, Faigenbaum AD, Stone MH, Oliver JL, Jeffreys I, Moody JA, Brewer C, Pierce KC, McCambridge TM, Howard R, Herrington L, Hainline B, Micheli LJ, Jaques R, Kraemer WJ, McBride MG, Best TM, Chu DA, Alvar BA, Myer GD. Position statement on youth resistance training: the 2014 International Consensus. Br J Sports Med. 2014 Apr;48(7):498-505. doi: 10.1136/bjsports-2013-092952. Epub 2013 Sep 20. PMID 24055781
- [Background] Malina RM. Weight training in youth-growth, maturation, and safety: an evidence-based review. Clin J Sport Med. 2006 Nov;16(6):478-87. doi: 10.1097/01.jsm.0000248843.31874.be. PMID 17119361
- [Background] Mazzulla M, Hodson N, West DWD, Kumbhare DA, Moore DR. A non-invasive 13CO2 breath test detects differences in anabolic sensitivity with feeding and heavy resistance exercise in healthy young males: a randomized control trial. Appl Physiol Nutr Metab. 2022 Aug 1;47(8):860-870. doi: 10.1139/apnm-2021-0808. Epub 2022 May 24. PMID 35609328
- [Background] Mazzulla M, Volterman KA, Packer JE, Wooding DJ, Brooks JC, Kato H, Moore DR. Whole-body net protein balance plateaus in response to increasing protein intakes during post-exercise recovery in adults and adolescents. Nutr Metab (Lond). 2018 Sep 24;15:62. doi: 10.1186/s12986-018-0301-z. eCollection 2018. PMID 30258470
- [Background] McKinlay BJ, Wallace P, Dotan R, Long D, Tokuno C, Gabriel DA, Falk B. Effects of Plyometric and Resistance Training on Muscle Strength, Explosiveness, and Neuromuscular Function in Young Adolescent Soccer Players. J Strength Cond Res. 2018 Nov;32(11):3039-3050. doi: 10.1519/JSC.0000000000002428. PMID 29337833
- [Background] Mersch, F., Stoboy, H., 1989. Strength training and muscle hypertrophy in children, in: Oseid, S., Carlsen, K. (Eds.), Children and Exercise XIII. Human Kinetics, Champaign, IL, pp. 165-182.
- [Background] Moore DR, Volterman KA, Obeid J, Offord EA, Timmons BW. Postexercise protein ingestion increases whole body net protein balance in healthy children. J Appl Physiol (1985). 2014 Dec 15;117(12):1493-501. doi: 10.1152/japplphysiol.00224.2014. Epub 2014 Oct 23. PMID 25342704
- [Background] Evans WJ, Shankaran M, Smith EC, Morris C, Nyangau E, Bizieff A, Matthews M, Mohamed H, Hellerstein M. Profoundly lower muscle mass and rate of contractile protein synthesis in boys with Duchenne muscular dystrophy. J Physiol. 2021 Dec;599(23):5215-5227. doi: 10.1113/JP282227. Epub 2021 Oct 11. PMID 34569076
- [Background] Schoenfeld, B., Fisher, J., Grgic, J., Haun, C., Helms, E., Phillips, S., Steele, J., Vigotsky, A., 2021. Resistance Training Recommendations to Maximize Muscle Hypertrophy in an Athletic Population: Position Stand of the IUSCA. International Journal of Strength and Conditioning 1, 1-30. https://doi.org/10.47206/ijsc.v1i1.81